CLINICAL TRIAL: NCT01090102
Title: Mesalamine to Reduce T Cell Activation in HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California HIV/AIDS Research Program (Other); Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 164320
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Immune System Diseases; Lentivirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Immune System Diseases; Lentivirus Infections; Acquired Immunodeficiency Syndrome | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Mesalamine (Experimental)
  Interventions: Drug: Mesalamine (5-aminosalicylic acid, Apriso)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesalamine (5-aminosalicylic acid, Apriso) — Four mesalamine capsules once daily (1.5 gram/day) for the first 12 weeks, PO(by mouth).
  Four placebo capsules once daily (1.5g/d) for another 12 weeks, PO (by mouth).
  Arms: Mesalamine
Drug: Placebo — Four placebo capsules once daily (1.5g/d) for the first 12 weeks, PO (by mouth).
  Four mesalamine capsules once daily (1.5g/d) for another 12 weeks, PO (by mouth).
  Arms: Placebo

SUMMARY:
The objective of this study is to determine whether 12 weeks of mesalamine therapy added to a standard HIV treatment decreases systemic immune activation and inflammation in HIV-infected patients, possibly resulting in better recovery of the immune system. The study hypothesis is that decreasing inflammation directly in the gut may decrease both of these potential causes of chronic inflammation, potentially resulting in an immunologic benefit.

DETAILED DESCRIPTION:
While most HIV-infected patients can now achieve nearly complete viral suppression on currently available HIV medications, they still have at least a 10-year shorter life expectancy than the general population and are at higher risk for diseases associated with accelerated aging including cardiovascular disease and non-AIDS-defining cancers. Persistent inflammation and immune activation are believed to drive this increased risk. Despite suppression of viral replication in peripheral blood by effective HIV medications, HIV may continue to be expressed at low levels by T cells in the lining of the gut and may also result in translocation of bacterial products across the lining of the gut, driving persistent inflammation. We believe that decreasing inflammation directly in the gut may decrease both of these potential causes of chronic inflammation, potentially resulting in an immunologic benefit. Mesalamine is an oral anti-inflammatory drug used to treat patients with inflammatory bowel disease, acts locally on the gut tissue to decrease inflammation, and is associated with very few side effects. If mesalamine therapy reduces immune activation and inflammation in our study, it would prompt larger studies to see if mesalamine decreases clinical outcomes like cardiovascular disease, cancer, and mortality in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry.
2. Stable antiretroviral therapy for at least 6 months.
3. Screening CD4+ T cell count below 350 cells/mm3
4. All available CD4+ T cell counts in the last year and at screening <350 cells/mm3
5. Screening plasma HIV RNA levels below level of detection (< 40 copies RNA/mL).
6. All available plasma HIV RNA levels within past year below the level of detection. Isolated detectable values < 500 c/ml are allowed if HIV RNA levels before and after this time point are undetectable.
7. >90% adherence to therapy within the preceding 30 days, as determined by self-report.
8. Both male and female subjects are eligible. Females of childbearing potential must have negative pregnancy test at screening and agree to use a double-barrier method of contraception during the study.

Exclusion Criteria:

1. Patients who are intending to modify antiretroviral therapy in the next 24 weeks for any reason.
2. Serious illness requiring hospitalization or parental antibiotics within preceding 3 months.
3. Exposure to any immunomodulatory drug in the past 16 weeks.
4. Active hepatitis C or hepatitis B which will require treatment in the subsequent 24 weeks.
5. Screening absolute neutrophil count <1,000 cells/mm3, platelet count <50,000 cells/mm3, Hgb < 8mg/dL
6. Pancreatitis or lipase greater than 2 times the upper limit of normal.
7. Renal insufficiency with creatinine clearance less than 50 ml/min
8. Elevated transaminases greater than 2.5 times the upper limit of normal.
9. Evidence of decompensated cirrhosis, heart failure.
10. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco-San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Somsouk M, Dunham RM, Cohen M, Albright R, Abdel-Mohsen M, Liegler T, Lifson J, Piatak M, Gorelick R, Huang Y, Wu Y, Hsue PY, Martin JN, Deeks SG, McCune JM, Hunt PW. The immunologic effects of mesalamine in treated HIV-infected individuals with incomplete CD4+ T cell recovery: a randomized crossover trial. PLoS One. 2014 Dec 29;9(12):e116306. doi: 10.1371/journal.pone.0116306. eCollection 2014. PMID 25545673

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesalamine Then Placebo: Mesalamine (5-aminosalicylic acid, Apriso): Four mesalamine capsules once daily (1.5 gram/day) for the first 12 weeks, PO(by mouth), followed by Four placebo capsules once daily (1.5g/d) for another 12 weeks, PO (by mouth).
- Placebo Then Mesalamine: Placebo: Four placebo capsules once daily (1.5g/d) for the first 12 weeks, PO (by mouth), followed by Four mesalamine capsules once daily (1.5g/d) for another 12 weeks, PO (by mouth).
Period: First 12 Weeks
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Started | 15 | 18
Completed | 11 | 16
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 1
Period: Second 12 Weeks
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Started | 11 | 16
Completed | 11 | 15
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [49 to 62] | 60 [49 to 62] | 55 [49 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Log(10) Change in % Activated (CD38+HLA-DR+)CD8+ T Cells During the First 12 Weeks of Study
Time Frame: Week 0, Week 12
Population: 1 participant assigned to first receive Mesalamine was excluded from analysis due to having withdrawn participation without receiving the allocated intervention
Measure: Mean (95% Confidence Interval); unit: Log10(percentage of T cells)
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Number analyzed (Participants) | 14 | 18
Log10(percentage of T cells) | 0.03 [-0.14 to 0.20] | -0.01 [-0.10 to 0.07]
Statistical Analysis 1: Comparison: Mesalamine Then Placebo vs Placebo Then Mesalamine; Test type: Superiority or Other; p = 0.63, t-test, 2 sided — Significant at p<0.05

2. Secondary Outcome: Log(10) Change in % Activated (CD38+HLA-DR+)CD8+ T Cells After Treatment Crossover
Description: Log(10) change in the percentage of activated T cells during the second 12 weeks of the study
Time Frame: Week 12, Week 24
Measure: Mean (95% Confidence Interval); unit: Log10(percentage of T cells)
Arm/Group | Mesalamine Then Placebo | Placebo Then Mesalamine
Number analyzed (Participants) | 11 | 16
Log10(percentage of T cells) | 0.003 [-0.19 to 0.19] | -0.03 [-0.15 to 0.08]
Statistical Analysis 1: Comparison: Mesalamine Then Placebo vs Placebo Then Mesalamine; Test type: Superiority or Other; p = 0.77, t-test, 2 sided — significant at p<0.05

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Mesalamine: Mesalamine (5-aminosalicylic acid, Apriso): Four mesalamine capsules once daily (1.5 gram/day) PO(by mouth).
- Placebo: Placebo: Four placebo capsules once daily (1.5g/d) PO (by mouth).
Arm/Group | Mesalamine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/29
Other Adverse Events (participants affected / at risk) | 2/31 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mesalamine (N=31) | Placebo (N=29)
Death (General disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mesalamine (N=31) | Placebo (N=29)
Liver Cirrhosis (Hepatobiliary disorders) | 1 | 0
Drug relapse (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes